CLINICAL TRIAL: NCT00747110
Title: Double-blind, Double-dummy, Randomised, Multi-centre, Comparative Phase III Clinical Study on the Efficacy and Tolerability of an 8 Week Oral Treatment With 9 mg Budesonide or 3 g Mesalazine in Patients With Active Ulcerative Colitis
Brief Title: Budesonide Capsules Versus Mesalazine Granules in Active Ulcerative Colitis (UC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUC-57/UCA; 2006-005377-22 (EudraCT Number)
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Colitis, Ulcerative
Keywords: 5-ASA; mesalamine; mesalazine; budesonide; ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Budesonide; Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): 9mg budesonide OD
  Interventions: Drug: budesonide
- B (Active Comparator): 3g mesalazine OD
  Interventions: Drug: mesalazine

INTERVENTIONS:
Drug: budesonide — 3x 3mg budesonide capsules once daily
  Other Names: Budenofalk 3mg capsules
  Arms: A
Drug: mesalazine — 3x 1000mg mesalazine onc daily
  Other Names: Salofalk 1000mg granules
  Arms: B

SUMMARY:
The purpose of this study is to prove the therapeutic equivalence and safety of once-daily 9 mg budesonide versus 3 g mesalazine in a 8-week treatment in patients with active ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent,
2. Men or women aged 18 to 75 years,
3. Active ulcerative colitis, except proctitis limited to 15 cm ab ano, confirmed by endoscopy and histology,
4. Established disease (presence of blood or mucus in the stools) or new diagnosis (bloody stools occurring at least during 14 days prior to baseline visit),
5. Clinical Activity Index (CAI) >= 6 and Endoscopical Index (EI) >= 4,
6. Women of child-bearing potential, if heterosexually active, have to apply a highly effective method of birth control, which is defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptive method, some intrauterine devices (IUDs), sexual abstinence, or vasectomised partner. The investigator is responsible for determining whether the subject has adequate birth control for study participation.

Exclusion Criteria:

1. Crohn's disease, indeterminate colitis, ischaemic colitis, radiation colitis, microscopic colitis (i.e., collagenous colitis and lymphocytic colitis),
2. Toxic megacolon,
3. Baseline stool positive for germs causing bowel disease,
4. Diarrhoea as a result of the presence of other symptomatic organic disease(s) of the gastrointestinal tract,
5. Active peptic ulcer disease,
6. Haemorrhagic diathesis,
7. Asthma, diabetes mellitus, infection, osteoporosis, glaucoma, cataract, or cardiovascular disease if careful medical monitoring is not ensured,
8. Severe co-morbidity substantially reducing life expectancy,
9. Active colorectal cancer or a history of colorectal cancer,
10. Active malignancy other than colorectal cancer or treatment with anticancer drugs during the last 5 years. Patients with a history of cancer other than colorectal cancer and at least five years of uneventful follow up and no signs of recurrence may be eligible,
11. Immunosuppressants within 3 months and/or corticosteroids (oral, intravenous [IV] or topical rectal) within 4 weeks prior to baseline,
12. Current relapse occurred under maintenance treatment with > 2.4 g mesalazine per day,
13. Abnormal renal function (Serum Cystatin C > upper limit of normal [ULN]),
14. Abnormal hepatic function (ALT, AST or AP >= 2 x ULN) or liver cirrhosis,
15. Known intolerance/hypersensitivity/resistance to study drugs or drugs of similar chemical structure or pharmacological profile, or to any of the other constituents of the study drugs,
16. Doubt about the patient's cooperation, e.g., because of addiction to alcohol or drugs,
17. Existing or intended pregnancy or breast-feeding,
18. Participation in another clinical trial within the last 30 days, simultaneous participation in another clinical trial, or previous participation in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2007-10; Primary Completion 2008-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Rate of clinical remission (defined by CAI <= 4, with stool frequency and rectal bleeding subscores of ´0´) at week 8 (LOCF) | week 8 (LOCF)

SECONDARY OUTCOMES:
Time to first resolution of clinical symptoms | within 8 weeks
CAI in the course of the study | week 0, 2, 4, 6, 8
Disease Activity Index (DAI)in the course of the study | week 0 and 8 (LOCF)
Endoscopical Index (EI)in the course of the study | week 0 and 8 (LOCF)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Mueller, Dr, Study Director — Dr. Falk Pharma GmbH
Locations (1):
- Klinikum St. Marien, Amberg, Germany

REFERENCES:
- [Result] Gross V, Bunganic I, Belousova EA, Mikhailova TL, Kupcinskas L, Kiudelis G, Tulassay Z, Gabalec L, Dorofeyev AE, Derova J, Dilger K, Greinwald R, Mueller R; International BUC-57 Study Group. 3g mesalazine granules are superior to 9mg budesonide for achieving remission in active ulcerative colitis: a double-blind, double-dummy, randomised trial. J Crohns Colitis. 2011 Apr;5(2):129-38. doi: 10.1016/j.crohns.2010.11.006. Epub 2010 Dec 14. PMID 21453882